CLINICAL TRIAL: NCT02171650
Title: A Phase I Open-label Extension Study of 1200.1 and 1200.2 of Once-daily Oral Treatment With BIBW 2992 in Patients With Advanced Solid Tumors
Brief Title: BIBW 2992 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.17
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Afatinib

ARMS (1):
- BIBW 2992 (Experimental)
  Interventions: Drug: BIBW 2992

INTERVENTIONS:
Drug: BIBW 2992

SUMMARY:
The primary objective was to collect safety data for BIBW 2992.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who have completed the prescribed courses of the 1200.1 or 1200.2 studies without clinical disease progression
* Age 18 years or older
* Life expectancy of at least three (3) months
* Written informed consent that is consistent with International Conference on Harmonization - Good Clinical Practice guidelines
* Eastern Cooperative Oncology Group (ECOG) performance score 0, 1 or 2
* Patients must be recovered from previous surgery

Exclusion Criteria:

* Active infectious disease
* Gastrointestinal disorders that may interfere with the absorption of the study drug or chronic diarrhea
* Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol
* Patients with untreated or symptomatic brain metastases. Patients with treated, asymptomatic brain metastases are eligible if there has been no change in brain disease status for at least eight (8) weeks, no history of cerebral edema or bleeding in the past eight (8) weeks and no requirement for steroids or anti-epileptic therapy
* Cardiac left ventricular function with resting ejection fraction >= CTC Grade 1
* Absolute neutrophil count (ANC) less than 1500 / mm3
* Platelet count less than 100 000 / mm3
* Bilirubin greater than 1.5 mg / dl (> 26 μmol / L, Systeme International (SI) unit equivalent)
* Aspartate amino transferase (AST) or alanine amino transferase (ALT) greater than three times the upper limit of normal (if related to liver metastases greater than five times the upper limit of normal)
* Serum creatinine greater than 1.5 mg / dl (> 132 μmol / L, SI unit equivalent)
* Women and men who are sexually active and unwilling to use a medically acceptable method of birth control
* Pregnancy or breast-feeding
* Treatment with other investigational drugs; chemotherapy, immunotherapy, radiotherapy or hormone therapy (excluding Luteinizing hormone-releasing hormone agonists, or other hormones taken for breast cancer, or bisphosphonates), or participation in a clinical study other than 1200.1 or 1200.2
* Patients unable to comply with the protocol
* Active alcohol or drug abuse
* Patients not recovered from any dose-limiting toxicity

The patients are eligible for re-treatment after the previous course is finished. Patients will not be eligible if the following conditions are met:

* Patients with clinical signs of disease progression or if latest X-ray, CT, MRI or US reveals progressive disease
* Cardiac left ventricular function CTC Grade ≥ 2 at any time during the previous course
* Patients fulfilling any of the Exclusion Criteria listed in Section 3.3 on Day 29 of the previous course
* Patient not recovered from any dose-limiting toxicity (DLT) 14 days after the last administration of BIBW2992 in the previous course. Recovery is defined as return to baseline condition (Visit 1 of 1200.1 or Visit 1 of 1200.2) or CTC Grade 1, whichever is higher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2004-12-01 (Actual); Primary Completion 2006-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events, according to Common Terminology Criteria (CTC) version 3, with particular scrutiny of events that were considered to be dose-limiting toxicities and those that were serious or significant | up to 18 months

SECONDARY OUTCOMES:
Durability of non-progression as measured by tumor assessment according to Response Evaluation Criteria in Solid Tumors (RECIST) | every 8 weeks up to 18 months

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com